CLINICAL TRIAL: NCT05059990
Title: Comparison of Low Intensity Aerobic Exercise and Active Exercises on Cancer Related Fatigue in Cancer Patients Receiving Palliative Care
Brief Title: Low Intensity Aerobic Exercise and Active Exercises in Cancer Patients Receiving Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REC/01085 Ishrat Perveen
Record Dates: First submitted 2021-09-18; First posted 2021-09-28 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Cancer
Keywords: Low intensity Aerobic Exercise; ROM Exercise; Palliative Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Intensity Aerobic Exercises Group (Experimental): stationary cycle for aerobic exercise
  Interventions: Other: Low Intensity Aerobic Exercises Group
- Active Exercises Group (Active Comparator): Upper and lower limb range of Motion (ROM) & stretching exercises uses in active exercise group
  Interventions: Other: Active Exercises Group

INTERVENTIONS:
Other: Low Intensity Aerobic Exercises Group — Intervention Low Intensity Aerobic Exercises i.e. stationary cycle(supervised) Intensity 55-65% of HRmax Frequency 3 times a week Duration 30 min each session
  Arms: Low Intensity Aerobic Exercises Group
Other: Active Exercises Group — Intervention Upper and lower limb ROM & stretching exercises Intensity As per tolerance Frequency 12 repetition/4sets per exercise 3 times/week Duration 30 minutes each session
  Arms: Active Exercises Group

SUMMARY:
To compare the effect of low intensity aerobic exercise and active ROM exercises on cancer related fatigue and its associated symptoms and quality of life in cancer patients receiving palliative care.

ELIGIBILITY:
Inclusion Criteria:

* ability to give written consent.
* Diagnosed advance cancer specifically gastrointestinal tract (GIT) cancer, Lung cancer and Breast cancer etc. (stage 2 and 3).
* Intensity of fatigue ≥4 out of 10 on fatigue Numerical Rating Scale in first visit observation
* Survival expectancy more than one month,
* Functional status allowing the participants to participate in the proposed therapy.

Exclusion Criteria:

* Anemia (Hb ≤ 8g/dl),
* Existence of other comorbidities causing fatigue (i.e. Parkinson's, Multiple sclerosis, Heart failure),
* Infection requiring antibodies
* bone metastases,
* thrombocytopenia (<50×109/l),
* myocardial infarction within the past three months
* uncontrolled hypertension (diastolic pressure >95 mm Hg).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Fatigue Numeric Rating Scale | 4th Week
  The fatigue numeric rating scale (NRS) is a single-item measure assessing severity of fatigue. We will use this in our study to measure the severity of cancer related fatigue in oncology patients receiving palliative care. The fatigue NRS is a patient- administered, single- item, 11- point horizontal scale anchored at 0 and 10, with 0 representing 'no fatigue' and 10 representing 'as bad as participant can imagine'. Changes from the baseline to 4 week
Karnofsky Performance Status | 4 Week
  The Karnofsky Performance Scale Index is an assessment tool for functional impairment. It can be used to compare effectiveness of different therapies and to assess the prognosis in individual patients. It is a standard way of measuring the ability of cancer patients to perform ordinary tasks. The Karnofsky Performance Status scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities. Changes from the baseline to 4 week
Edmonton Symptom Assessment Scale (ESAS) | 4 week
  This tool is designed to assess nine common symptoms experienced by cancer patients, including pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, shortness of breath. The severity for each symptom ranges from 0 to 10 where 0 means absence of symptom to 10 being the worst possible severity. Changes from the baseline to 4 week
Brief Fatigue Inventory (BFI): | 4 week
  It is used to rapidly assess the severity and impact of cancer-related fatigue on daily functioning in past 24 hours, which requires a very short time to fill and the global fatigue scoring can be obtained by averaging all the 4 items on the BFI. Changes from the baseline to 4 week

SECONDARY OUTCOMES:
Quality of life questionnaire for cancer patients treated with anti-cancer drugs (QOL-ACD): | 4 week
  Quality of Life Anti-Cancer Drugs (QOL-ACD) is a Quality-of-life measurement tool for patients undergoing chemotherapy it has 22 items, divided into these categories: daily activities, physical condition, social activities, mental and psychological status. Scaling of items is from 5 to 1(5 being worst and 1 being good) for 21 items, and a five-point face scale for 1 item. Changes from the baseline to 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University; Abeer Fatima, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Mubarak Hospital, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No